CLINICAL TRIAL: NCT06631677
Title: An Open Label, Expanded Access Program of Dupilumab in Adults With Severe IgE-Mediated Food Allergy Who Have Been Previously Treated With Linvoseltamab and Background Dupilumab
Brief Title: Expanded Access Program of Dupilumab in Adults With Severe Immunoglobulin E (IgE)-Mediated Food Allergy Who Have Been Previously Treated With Linvoseltamab and Background Dupilumab in the Parent Study R5458-668-ALG-2219 (NCT06369467)
Status: No longer available | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R668-ALG-2448
Record Dates: First submitted 2024-09-19; First posted 2024-10-08 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — dupilumab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Dupilumab — Administered per protocol
  Other Names: REGN668; DUPIXENT®; SAR231893

SUMMARY:
This is an expanded access program of dupilumab that was never initiated and, therefore, not available.

Age Groups: Child, Adult, Older Adult